CLINICAL TRIAL: NCT04738032
Title: Stories for Change: Digital Storytelling Intervention for Diabetes Self-Management in the COVID-19 Pandemic
Acronym: S4C - COVID-19
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Hennepin Healthcare Research Institute (Other); Mountain Park Health Center (Unknown)
Responsible Party: Principal Investigator, Mark L Wieland, Mark Wieland, MD, MPH, Mayo Clinic
Other Study IDs: 20-006354
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Digital Storytelling Intervention — 12-minute digital storytelling intervention in Spanish, with four individuals explaining their personal Type 2 Diabetes stories.

SUMMARY:
Hispanic adults are twice as likely to have type 2 diabetes mellitus (T2D) and 1.5 times more likely to die from the disease than non-Hispanic whites. These disparities are mediated, in part, by less healthful levels of physical activity, dietary quality, medication adherence, and self-monitoring of blood glucose than non-Hispanic whites. Innovative approaches that arise from affected communities are needed to address these health disparities.

Community-based participatory research (CBPR) has been successful in targeting health issues among Hispanic and immigrant populations; CBPR is an effective approach for addressing health behaviors in a sociocultural context. In 2004, the research team developed a CBPR partnership between immigrant communities and academic institutions called Rochester Healthy Community Partnership (RHCP)

Storytelling or narrative-based interventions are designed to incorporate culture-centric health messaging to promote behavior change among vulnerable populations. Digital storytelling interventions are narrative-based videos elicited through a CBPR approach to surface the authentic voices of individuals overcoming obstacles toward engaging in health promoting behaviors to shape positive health behaviors of viewers through influences on attitudes and beliefs.

RHCP partners from Hispanic communities identified T2D as a priority area for intervention, and have co-created each of the formative phases leading up to this proposal. Narrative theory and social cognitive theory formed the conceptual basis for intervention development. The study team conducted surveys and focus groups to derive the approach and personnel for building an authentic intervention that was created in a digital storytelling workshop where stories about diabetes self-management were captured, recorded, and edited to derive the final intervention products in video forma. The respective digital storytelling videos were pilot tested with 25 patients across healthcare institutions in Minnesota and Arizona. The intervention was rated as highly acceptable, culturally relevant, and perceived as efficacious for motivating behavioral change.

The overall objective of this project is therefore to assess the efficacy of a digital storytelling intervention derived through a CBPR approach on self-management of T2D among Hispanic adults during a pandemic.

DETAILED DESCRIPTION:
The study team will conduct an observational trial in a virtual settings at two healthcare institutions among 80 Hispanic adults with poorly controlled T2D (hemoglobin A1c≥8%) who participated in a parent study, but were previously randomized to the Control group. The participants will view the 12-minute digital storytelling video, as well as completed a brief survey regarding how the pandemic may have affected their diabetes self-care.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Hispanic or Latino.
* Between 18 and 70 years of age.
* Participated in the parent study

Exclusion Criteria:

* Does not self-identifies as Hispanic or Latino.
* Is not between 18 and 70 years of age.
* Did not participated in the parent study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Self-identifies as Hispanic or Latino and has poorly controlled type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Diabetes self-management behaviors | 5 months
  This is a brief survey instrument to assess the following domains: general diet, specific (diabetes) diet, physical activity, diabetes medication use, and blood glucose monitoring during the pandemic.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mountain Park Health Center, Phoenix, Arizona
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No